CLINICAL TRIAL: NCT05911295
Title: An Open-label, Randomized, Controlled Phase 3 Study of Disitamab Vedotin in Combination With Pembrolizumab Versus Chemotherapy in Subjects With Previously Untreated Locally Advanced or Metastatic Urothelial Carcinoma That Expresses HER2 (IHC 1+ and Greater)
Brief Title: Disitamab Vedotin With Pembrolizumab vs Chemotherapy in Previously Untreated Urothelial Cancer Expressing HER2
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Seagen, a wholly owned subsidiary of Pfizer (Industry)
Collaborators: RemeGen Co., Ltd. (Industry); Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Organization: Seagen Inc. (Industry)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SGNDV-001; C5731001 (Other: Alias Study Number); 2022-501105-12-00 (Registry Identifier: CTIS (EU))
Record Dates: First submitted 2023-06-09; First posted 2023-06-22 (Actual); Last update posted 2025-12-15 (Actual); Status verified 2025-12

CONDITIONS: Urothelial Carcinoma
Keywords: Urothelial Cancer; LA/mUC; Bladder Cancer; HER2 Overexpression; HER2 Amplification; HER2; Seattle Genetics
MeSH Terms: conditions — Carcinoma, Transitional Cell; Urinary Bladder Neoplasms | interventions — disitamab vedotin; RC48 antibody; pembrolizumab; Gemcitabine; Cisplatin; Carboplatin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Disitamab vedotin arm (Experimental): disitamab vedotin + pembrolizumab
  Interventions: Drug: disitamab vedotin; Drug: pembrolizumab
- Standard of care arm (Active Comparator): gemcitabine + cisplatin OR carboplatin
  Interventions: Drug: gemcitabine; Drug: cisplatin; Drug: carboplatin

INTERVENTIONS:
Drug: disitamab vedotin — Given into the vein (IV; intravenous) every 2 weeks
  Other Names: RC48, RC48-ADC
  Arms: Disitamab vedotin arm
Drug: pembrolizumab — 400mg given by IV every 6 weeks
  Other Names: KEYTRUDA®
  Arms: Disitamab vedotin arm
Drug: gemcitabine — 1000 mg/m^2 given by IV on days 1 and 8 of every 3-week cycle
  Other Names: Gemzar
  Arms: Standard of care arm
Drug: cisplatin — 70 mg^2 given by IV on day 1 of every 3-week cycle
  Arms: Standard of care arm
Drug: carboplatin — Area under the plasma concentration-time curve (AUC) 4.5 or 5 given by IV on day 1 of every 3-week cycle
  Arms: Standard of care arm

SUMMARY:
This study will enroll participants with urothelial cancer (UC). UC can include cancer of the bladder, kidney, or the tubes that carry pee through the body (ureter, urethra). This study will try to find out if the drugs disitamab vedotin with pembrolizumab works better than platinum-containing chemotherapy to treat patients with UC. This study will also test what side effects happen when participants take these drugs together. A side effect is anything a drug does to the body besides treating the disease.

Participants in this study will have cancer that has spread through the body (metastatic) or spread near where it started (locally advanced).

In this study, there are 2 different groups. Participants will be assigned to a group randomly. Participants in the disitamab vedotin arm will get the study drug disitamab vedotin once every two weeks and pembrolizumab once every 6 weeks. Participants in the standard of care arm will get gemcitabine once a week for 2 weeks with either cisplatin or carboplatin once every 3 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Histopathological confirmation of locally advanced unresectable or metastatic urothelial carcinoma (LA/mUC), including UC originating from the renal pelvis, ureters, bladder, or urethra.
* Measurable disease by investigator assessment per RECIST v1.1.
* Participant must not have received prior systemic therapy for LA/mUC. Exception will be made for neoadjuvant or adjuvant therapy, if disease recurrence/progression occurred more than 12 months after the last dose of therapy.
* Eligible to receive cisplatin- or carboplatin-containing chemotherapy.
* Able to provide archived formalin-fixed paraffin-embedded tumor tissue blocks from a muscle-invasive or metastatic UC lesion or biopsy of metastatic UC prior to treatment initiation. If archival tissue is not available a newly obtained baseline biopsy of an accessible tumor lesion is required within 28 days of cycle 1 day 1.
* HER2 expression of 1+ or greater on immunohistochemistry (IHC).
* Eastern Cooperative Oncology Group (ECOG) performance score of 0, 1, or 2 within 7 days prior to randomization.

Exclusion Criteria:

* Known hypersensitivity to disitamab vedotin, cisplatin, carboplatin, gemcitabine, or pembrolizumab or any of their components.
* History of severe/life threatening immune-related adverse event (irAE) with PD-(L)1 inhibitors are excluded.
* Central nervous system (CNS) and/or leptomeningeal metastasis. Participants with treated CNS metastases are permitted if all of the following are met.

  * CNS metastases have been clinically stable for at least 4 weeks and baseline scans show no evidence of new or worsening CNS metastasis.
  * Participant is on a stable dose of ≤ 10 mg/day of prednisone or equivalent for at least 2 weeks.
* History of or active autoimmune disease that has required systemic treatment in the past 2 years.
* Prior treatment with an agent directed to another stimulatory or co-inhibitory T cell receptor (including but not limited to CD137 agonists, CAR-T cell therapy, CTLA-4 inhibitors, or OX-40 agonists).
* Prior solid organ or bone marrow transplantation.
* Pleural effusion or ascites with symptoms or requiring symptomatic treatment.
* Estimated life expectancy <12 week
* Prior treatment with an MMAE agent or anti-HER2 therapy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 400 (Estimated)
Dates: Start 2023-09-22 (Actual); Primary Completion 2026-06-30 (Estimated); Study Completion 2029-04-30 (Estimated)

PRIMARY OUTCOMES:
Progression-free survival (PFS) per Response Evaluation Criteria in Solid Tumors version 1.1 (RECIST v1.1) by blinded independent central review (BICR) | Approximately 3 years
  The time from randomization to first documentation of disease progression per RECIST v1.1 by BICR, or to death due to any cause.
Overall survival (OS) | Approximately 5 years
  The time from date of randomization to date of death due to any cause.

SECONDARY OUTCOMES:
Objective response rate (ORR) per RECIST v1.1 by BICR | Approximately 3 years
  The proportion of participants with confirmed complete response (CR) or partial response (PR) according to RECIST v1.1.
ORR per RECIST v1.1 by investigator assessment | Approximately 3 years
  The proportion of participants with confirmed CR or PR according to RECIST v1.1.
Duration of Response (DOR) per RECIST v1.1 by BICR | Approximately 3 years
  The time from first documented response of CR or PR (that is subsequently confirmed) to the first documented disease progression per RECIST v1.1, or to death due to any cause.
DOR per RECIST v1.1 by investigator assessment | Approximately 3 years
  The time from first documented response of CR or PR (that is subsequently confirmed) to the first documented disease progression per RECIST v1.1, or to death due to any cause.
Control Rate (DCR) per RECIST v1.1 by BICR | Approximately 3 years
  The proportion of participants with confirmed CR, PR, or stable disease according to RECIST v1.1.
DCR per RECIST v1.1 by investigator assessment | Approximately 3 years
  The proportion of participants with confirmed CR, PR, or stable disease according to RECIST v1.1.
PFS per RECIST v1.1 by investigator assessment | Approximately 3 years
  The time from randomization to first documentation of disease progression per RECIST v1.1, or to death due to any cause.
Number of participants with adverse events (AEs) | Through 30 days after the last study treatment; approximately 2 years
  Any untoward medical occurrence in a clinical study participant, temporally associated with the use of study intervention, whether or not considered related to the study intervention.
Number of participants with laboratory abnormalities | Through 30 days after the last study treatment; approximately 2 years
Treatment discontinuation rate due to AEs | Approximately 2 years
Number of electrocardiogram (ECG) abnormalities | Through 30 days after the last study treatment; approximately 2 years
Change from baseline of left ventricular ejection fraction (LVEF) | Through 2 years after last study treatment; approximately 4 years
Change from baseline to Week 16 in European Organization for Research and Treatment of Cancer core Quality of Life questionnaire (EORTC QLQ-C30) Global Health Status (GHS)/QoL Score | Approximately 2 years
  The EORTC QLQ-C30 is used to evaluate health-related quality of life, functioning, disease symptoms, and treatment-related side effects. Scores range from 0-100. For GHS/QoL and functional scales, higher scores represent higher QoL or functioning. For symptom scales, higher scores represent more symptoms/worse status.
Time to Deterioration in EORTC QLQ-C30 GHS/QoL Score | Approximately 2 years
  The time from the date of randomization to the date of first deterioration (change from baseline ≥10) in GHS/QoL score with no subsequent recovery. The EORTC QLQ-C30 is used to evaluate health-related quality of life, functioning, disease symptoms, and treatment-related side effects. Scores range from 0-100. For GHS/QoL and functional scales, higher scores represent higher QoL or functioning. For symptom scales, higher scores represent more symptoms/worse status.
Time to pain progression | Approximately 2 years
  The time from the date of randomization to whichever of the following occurs earlier:
  * an increase in Numeric Rating Scale (NRS) for pain intensity of 2 points or more from baseline at 2 consecutive visits,
  * an increase in number of opioid or analgesic use from baseline,
  * or initiation of opioid or analgesic use. NRS for pain intensity asks participants to best describe their pain at its worst in the last 24 hours from 0 to 10. On the NRS, 0 means no pain and 10 means pain as bad as you can imagine.

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (347):
- United States (108):
  - Banner Gateway Medical Center, Gilbert, Arizona
  - Banner MD Anderson Cancer Center, Gilbert, Arizona
  - UCLA Hematology/Oncology - Alhambra, Alhambra, California
  - Foothill Cardioology, Arcadia, California
  - Beverly Hills Multi-Specialties Practice, Beverly Hills, California
  - Providence Saint Joseph Medical Center, Burbank, California
  - UCLA Burbank Cardiology, Burbank, California
  - UCLA Hematology/Oncology - Burbank, Burbank, California
  - UCLA Calabasas Specialty Care, Calabasas, California
  - UCLA Encino Specialty Care (Radiology), Encino, California
  - UCLA Hematology/Oncology - Encino, Encino, California
  - Helios Clinical Research, Fountain Valley, California
  - Helios Clinical Research, Glendale, California
  - Foothill Cardiology Glendora, Glendora, California
  - Helios Clinical Research, Long Beach, California
  - UCLA Downtown Los Angeles Primary & Specialty Care, Los Angeles, California
  - UCLA Cardiovascular Center, Los Angeles, California
  - UCLA Department of Medicine-Hematology/Oncology, Los Angeles, California
  - UCLA Hematology & Oncology Clinic, Los Angeles, California
  - UCLA Hematology / Oncology, Los Angeles, California
  - UCLA Westwood Specialty Care, Los Angeles, California
  - UCLA Montecito Primary & Specialty Care, Montecito, California
  - Pacific Cancer Care, Monterey, California
  - Newport Diagnostics, Newport Beach, California
  - Foothill Cardiology Pasadena, Pasadena, California
  - Southern California Heart Specialists, Pasadena, California
  - UCLA Porter Ranch Primary & Specialty Care, Porter Ranch, California
  - UCSF Center at China Basin Imaging, San Francisco, California
  - Helen Diller Family Comprehensive Cancer Center - Imaging Divisadero, San Francisco, California
  - Helen Diller Family Comprehensive Cancer Center - Imaging Post, San Francisco, California
  - UCSF Cancer Center MZ Phlebotomy, San Francisco, California
  - UCSF Helen Diller Family Comprehensive Cancer Center, San Francisco, California
  - UCSF Mount Zion Phlebotomy, San Francisco, California
  - UCSF Parnassus Phlebotomy, San Francisco, California
  - UCSF Parnassus-5 Lab, San Francisco, California
  - Cardiovascular Care and Prevention Center at Mission Bay, San Francisco, California
  - The Regents of the University of California, San Francisco, California
  - UCSF Investigational Drugs Pharmacy, San Francisco, California
  - UCSF Mission Bay Gateway-2 Lab, San Francisco, California
  - UCSF Mission Bay PCMB-5 Lab, San Francisco, California
  - UCSF Mission Bay Pediatric Clinical Research Center, San Francisco, California
  - UCSF Mission Bay Radiology and Nuclear Medicine, San Francisco, California
  - University of California San Francisco, San Francisco, California
  - University of California, San Francisco | HDFCCC - Hematopoietic malignancies, San Francisco, California
  - Diagnostic Medical Group of Southern California, , San Gabriel, CA, San Gabriel, California
  - Southern California Heart Centers, San Gabriel, California
  - UCLA Hematology/Oncology - San Luis Obispo, San Luis Obispo, California
  - Sierra Vista Regional Medical Center, San Luis Obispo, California
  - Helios Clinical Research, Santa Ana, California
  - UCLA Hematology/Oncology - Santa Barbara, Santa Barbara, California
  - UCLA Santa Monica Cardiology, Santa Monica, California
  - UCLA Simi Valley Alamo Specialty Care, Simi Valley, California
  - Twin Cities Community Hospital, Templeton, California
  - UCLA Thousand Oaks Primary & Specialty Care, Thousand Oaks, California
  - UCLA Hematology/Oncology - Torrance, Torrance, California
  - UCLA Torrance Lomita Specialty Care, Torrance, California
  - UCLA Santa Clarita Primary & Specialty Care, Valencia, California
  - UCLA Ventura Cardiology, Ventura, California
  - UCLA Hematology/Oncology - Westlake, Westlake Village, California
  - Helios Clinical Research, Whittier, California
  - Greater Baltimore Medical Center, Baltimore, Maryland
  - HealthPartners Institute, Bloomington, Minnesota
  - M Health Fairview Ridges Cancer Clinic, Burnsville, Minnesota
  - Minnesota Oncology Hematology, PA, Burnsville, Minnesota
  - Allina Health Cancer Institute, Coon Rapids, Minnesota
  - Minnesota Oncology Hematology, PA, Coon Rapids, Minnesota
  - M Health Fairview Cancer Clinic-Edina, Edina, Minnesota
  - Minnesota Oncology Hematology Pa, Edina, Minnesota
  - Minnesota Oncology Hematology, PA, Fridley, Minnesota
  - M Health Fairview Maple Grove Cancer Center, Maple Grove, Minnesota
  - Minnesota Oncology Hematology, PA, Maplewood, Minnesota
  - Allina Health Cancer Institute-United(VPCI), Minneapolis, Minnesota
  - Minnesota Oncology Hematology, PA, Minneapolis, Minnesota
  - Hennepin Country Medical Center, Minneapolis, Minnesota
  - M Health Fairview University of Minnesota Investigational Drug Services, Minneapolis, Minnesota
  - Metro Minnesota Community Oncology Research Consortium(MMCORC), Saint Louis Park, Minnesota
  - Regions Hospital, Saint Paul, Minnesota
  - Allina Health Cancer Institute-United(VPCI), Saint Paul, Minnesota
  - Minnesota Oncology Hematology, PA, Woodbury, Minnesota
  - M Health Fairview Lakes Medical Center, Wyoming, Minnesota
  - Nebraska Medicine- Bellevue Medical Center, Bellevue, Nebraska
  - Nebraska Medicine -Nebraska Medical Center, Omaha, Nebraska
  - Nebraska Medicine-Cancer Center at Village Pointe Health Center, Omaha, Nebraska
  - The University of Nebraska Medical Center, Omaha, Nebraska
  - University of Nebraska Medical Center, Omaha, Nebraska
  - Optum Care Cancer Care at Seven Hills, Las Vegas, Nevada
  - OptumCare Cancer center, Las Vegas, Nevada
  - Icahn School of Medicine at Mount Sinai, New York, New York
  - Ship study drug to: Mount Sinai Hospital- Pharmacy Dept, New York, New York
  - ECU Health Medical Center, Greenville, North Carolina
  - AHN Saint Vincent Hospital, Erie, Pennsylvania
  - AHN Jefferson Hospital, Jefferson Hills, Pennsylvania
  - AHN Forbes Hospital, Monroeville, Pennsylvania
  - Allegheny Valley Hospital, Natrona Heights, Pennsylvania
  - AHN Cancer Institute - Allegheny General Hospital, Pittsburgh, Pennsylvania
  - AHN Cancer Institute Pharmacy, Pittsburgh, Pennsylvania
  - AHN West Penn Hospital, Pittsburgh, Pennsylvania
  - University of Texas Southwestern Medical Center - Simmons Cancer Center, Dallas, Texas
  - UT Southwestern Medical Center - Redbird, Dallas, Texas
  - University of Texas Southwestern Medical Center-Simmons Cancer Center Pharmacy, Dallas, Texas
  - University of Texas Southwestern Medical Center, Dallas, Texas
  - UT Southwestern - Simmons Cancer Center - Fort Worth, Fort Worth, Texas
  - UT Southwestern - Simmons Cancer Center - Richardson/Plano, Richardson, Texas
  - Inova Schar Cancer Institue Infusion Pharmacy, Fairfax, Virginia
  - Inova Schar Cancer Institute, Fairfax, Virginia
  - Harborview Medical Center, Seattle, Washington
  - Fred Hutchinson Cancer Center., Seattle, Washington
  - University of Washington Medical Center, Seattle, Washington
- Argentina (22):
  - Centro de Investigacion Pergamino SA, Pergamino, Buenos Aires
  - Centro de Investigaciones Medicas y Desarrollo LC, Buenos Aires, Buenos Aires F.D.
  - Clinica Viedma, Viedma, Río Negro Province
  - Fundación Dr. Ruben Kowalyszyn, Viedma, Río Negro Province
  - Sanatorio Parque, Rosario, Santa Fe Province
  - Centro de Oncologia e Investigacion de Buenos Aires (COIBA), Berazategui
  - Labmedicina, Buenos Aires
  - Fundacion CENIT para la lnvestigacion en Neurociencias, Buenos Aires
  - Instituto Médico Especializado Alexander Fleming, Buenos Aires
  - Centro Oncologico Korben, Buenos Aires
  - Centro Medico Austral, Buenos Aire
  - Centro Oncologico Korben, Buenos Aire
  - Fundacion Cenit, CABA
  - Investigaciones Clinicas Moleculares (ICM), CABA
  - Clínica Universitaria Reina Fabiola, Córdoba
  - CEMAIC - Centro Medico Privado, Córdoba
  - Hospital Municipal de Morón. O. B. Lavignolle, Morón
  - Comité Provincial de Bioética-Rosario, Rosario
  - Grupo de Investigación en Oncología Clínica del Santario Parque, Rosario
  - Consultorio Dr. Miguel Angel Escudero, Salta
  - Oncologia Salta, Salta
  - Centro para la Atencion Integral del paciente Oncologico, San Miguel de Tucumán
- Australia (21):
  - Concord Repatriation General Hospital, Concord, New South Wales
  - Saint Vincents Hospital Sydney - Human Research Ethics Committee, Darlinghurst, New South Wales
  - St Vincent's Clinic, Darlinghurst, New South Wales
  - St George Hospital, Kogarah, New South Wales
  - Macquarie University Hospital, Macquarie University, New South Wales
  - Macquarie University, North Ryde, New South Wales
  - Prince of Wales Hospital, Randwick, New South Wales
  - North Shore Private Hospital, St Leonards, New South Wales
  - Mater Misericordiae - Mater Hospital Brisbane, Brisbane, Queensland
  - ICON Cancer Centre Chermside, Chermside, Queensland
  - Icon Cancer Centre Chermside, Herston, Queensland
  - Mater Research, South Bribane, Queensland
  - Peninsula & South Eastern Hematology and Oncology Group (PASO), Frankston, Victoria
  - Cabrini Hospital, Malvern, Victoria
  - Austin Health, Melbourne, Victoria
  - South Eastern Sydney Local Health District, Caringbah
  - Lyell McEwin Hospital, Elizabeth Vale
  - Peninsula And South East Oncology, Frankston
  - Mid North Coast Local Health District, NSW
  - Port Macquarie Base Hospital, Port Macquarie
  - Royal North Shore Hospital, St Leonards
- Belgium (5):
  - Algemeen Ziekenhuis Maria Middelares, Ghent
  - AZ St. Lucas, Ghent
  - University Hospital Ghent, Ghent
  - CHU de Liege Service Oncologie Medicale, Liège
  - CHU UCL Namur-Site de Saint Elisabeth, Namur
- Brazil (14):
  - Suporte Nutricional e Quimioterapia - PRONUTRIR, Fortaleza, Ceará
  - Centro de Oncologia da Bahia, Salvador, Estado de Bahia
  - Centro de Oncologia Hospital Sírio Libanês, Brasília, Federal District
  - Associacao Mario Penna - Hospital Luxemburgo - NEPI Nucleo de Ensino Pesquisa e Inovacao, Belo Horizonte, Minas Gerais
  - Hospital Sao Vicente de Paulo, Passo Fundo, Rio Grande do Sul
  - Hospital Mae de Deus, Porto Alegre, Rio Grande do Sul
  - Pontificia Universidade Catolica do Rio Grande do Sul (PUCRS), Porto Alegre, Rio Grande do Sul
  - Hospital Nossa Senhora da Conceicao / Grupo Hospitalar Conceicao, Porto Alegre, Rio Grande do Sul
  - Fundacao Doutor Amaral Carvalho, Jaú, São Paulo
  - Instituto de Ensino e Pesquisa - Sociedade Beneficente de Senhoras Hospital Sirio Libanes, São Paulo, São Paulo
  - Hospital de Cancer de Barretos - Fundacao Pio XII, Barretos
  - Erasto Gaertner Hospital, CuriBba
  - Instituto Nacional De Cancer - INCA, Rio de Janeiro
  - Hospital Alemao Oswaldo Cruz, São Paulo
- Canada (5):
  - Arthur J.E. Child Comprehensive Cancer Centre, Calgary, Alberta
  - University of Alberta / Cross Cancer Institute, Edmonton, Alberta
  - Lakeridge Health - The R.S. McLaughlin Durham Regional Cancer Centre (MDRCC), Oshawa, Ontario
  - University Health Network, Toronto, Ontario
  - Princess Margaret Cancer Centre - University Health Network, Toronto, Ontario
- Chile (7):
  - Centro de Oncologia de Precision, Los Condes, Region Metropolitana Santiago
  - Fundacion Arturo Lopez Perez, Providencia, Santiago Metropolitan
  - Oncovida - Santiago, Santiago, Santiago Metropolitan
  - Cesfar, Santiago, Santiago Metropolitan
  - Centro de Investigacion Clinica Bradford Hill, Santiago, Santiago Metropolitan
  - Centro de Estudios Clínicos SAGA, Santiago
  - Centro de Investigaciones Clinicas Vina del Mar, Viña del Mar
- Czechia (2):
  - Fakultni nemocnice Hradec Kralove, Hradec Králové, Hradec Králové
  - Fakultni Nemocnice Olomouc (Fnol) - Onkologicka Klinika, Olomouc
- France (8):
  - Centre Paul Strauss, Starsbourg, Grand Est
  - Hospices Civils de Lyon - Hopitale Lyon Sud, Pierre-Bénite, Rhône
  - University Hospital of Besancon, Besançon
  - Institut Bergonié Centre de Lutte Contre le Cancer (CLCC), Bordeaux
  - Polyclinique de Limoges Site Chenieux, Limoges
  - Unite de Coordination de la Biologie des Essais Cliniques, Strasbourg
  - Institut de Cancerologie Strasbourg Europe, Strasbourg
  - Institut Gustave Roussy, Villejuif
- Greece (3):
  - Athens Medical Center, Marousi, Attikí
  - Bioclinic Thessalonikis Private Clinic Single Member S.A., Thessaloniki, Kentrikí Makedonía
  - Metropolitan General Hospital, Cholargós
- Hungary (3):
  - Semmelweis Egyetem Urologiai Klinika, Budapest
  - Országos Onkológiai Intézet, Budapest
  - Bacs-Kiskun Varmegyei Oktatokorhaz, Kecskemét
- Ireland (5):
  - Cancer Trials Cork, Cork
  - Mater Misericordiae University Hospital, Dublin
  - Beaumont Hospital, Dublin
  - Tallaght University Hospital, Tallaght
  - Cork University Hospital, Wilton
- Israel (9):
  - Shaare Zedek Medical Center, Jerusalem, Other
  - Sheba Medical Center., Ramat Gan, Other
  - Emek Medical Center, Afula
  - Soroka Medical Center, Beersheba
  - Rambam Health Care Campus, Hafia
  - Hadassah University Hospital at Ein Kerem, Jerusalem
  - Meir Medical Center, Kefar Sava
  - Rabin Medical Center, Petah Tikva
  - Tel Aviv Sourasky Medical Center, Tel Aviv
- Italy (28):
  - IRCCS Istituto Tumori Giovanni Paolo II, Bari, Apulia
  - Azienda Ospedaliera Cardinale Giovanni Panico, Tricase, Apulia
  - IRCCS Istituto Romagnolo per lo Studio dei Tumori Dino Amadori- IRST S.r.l, Meldola (Fc), Emilia-Romagna
  - Ospedale Policlinico San Martino, Genoa, Liguria
  - Ospedale San Raffaele, Milan, Lombardy
  - IRCCS Istituto Clinico Humanitas, Rozzano, Milano
  - IRCCS San Raffaele Hospital ,Genitourinary medical Oncology, Lombardy, Milan
  - Azienda Sanitaria Locale Napoli 2 Nord, Giugliano in Campania, Naples
  - Azienda Ospedaliero-Universitaria Consorziale Policlinico di Bari, Bari, Other
  - P.O. "S. Maria Delle Grazie" - Pozzuoli - ASL Napoli Nord 2, Pozzuoli (NA), Other
  - SOSD Farmacia Ospedaliera, Aviano, Pordenone
  - Centro di Riferimento Oncologico Di Aviano, Aviano, Pordenone
  - AUSL Romagna - Presidio Ospedale "Umberto I" di Lugo, Lugo, Ravenna
  - AUSL della Romagna - Ospedale degli infermi, Faenza, RA
  - Fondazione Policlinico Agostino Gemelli IRCCS, Rome, ROMA
  - Azienda Ospedaliero Universitaria Careggi-SODc Oncologia Clinica (Padiglione16), Florence, Tuscany
  - ASST Cremona Farmacia Ospedaliera, Cremona
  - U.O. Farmacia Ospedaliera a Politiche del Farmaco Az. Osp. Universitaria Careggi, Florence
  - Ospedale Policlinico San Martino Farmacia, Genova
  - Istituto Nazionale Tumori IRCCS Fondazione G.Pascale Napoli Pascale, Napoli
  - SC Farmacia Ospedaliera C/O Istituto Nazionale Tumori IRCCS Fondazione G.Pascale Napoli Pascale, Napoli
  - Istituto Oncologico Veneto - IRCCS, Padua
  - Azienda Ospedaliera Universitaria Pisana Ospedale Santa Chiara, Pisa
  - Azienda Ospedaliera Universitaria Pisana, U.O. Farmacia Ospedaliera, Pisa
  - Unita Operative di Oncologia,Ospedale S.Maria delle Croci, Ravenna
  - SC ONCOLOGYA Medica e Traslazionale Azienda Ospedaliera S.Maria di terni, Terni
  - Azienda Ospedaliera Universitaria Integrata di Verona, Verona
  - Centro Ricerche Cliniche Di Verona Srl, Verona
- Japan (21):
  - Hirosaki University Hospital, Hirosaki, Aomori
  - Ehime University Hospital, Tōon, Ehime
  - National Hospital Organization Kyushu Cancer Center, Fukuoka, Fukuoka
  - Gunma Prefectural Cancer Center, Ota-Shi, Gunma
  - Kobe University Hospital, Kobe, Hyōgo
  - University of Tsukuba Hospital, Tsukuba, Ibaraki
  - Kagawa University Hospital, Kita-gun, Kagawa-ken
  - Yokohama City University Medical Center, Yokohama, Kanagawa
  - Kanagawa Cancer Center, Yokohama, Kanagawa
  - University of Miyazaki Hospital, Miyazaki, Miyazaki
  - Nara Medical University Hospital, Kashihara, Nara
  - Kindai University Hospital, Osakasayama-Shi, Osaka
  - Osaka University Hopsital, Suita, Osaka
  - Tokushima University Hospital, Tokushima, Tokushima
  - Keio University Hospital, Shinjuku-ku, Tokyo
  - Wakayama Medical University Hospital, Wakayama, Wakayama
  - Yamaguchi University Hospital, Ube, Yamaguchi
  - Chiba Cancer Center, Chiba
  - National Hospital Organization Kumamoto Medical Center, Kumamoto
  - Osaka Prefectural Hospital Organization - Osaka International Cancer Institute, Osaka
  - Yamagata University Hospital, Yamagata
- Netherlands (7):
  - Antoni van Leeuwenhoek Apotheek,I-2, Amsterdam
  - Netherlands Cancer Institute/Antoni van Leeuwenhoek, Amsterdam
  - Rijnstate Hospital, Arnhem
  - Amphia Ziekenhuis, Breda
  - Maastricht Universitair Medisch Centrum+, Maastricht
  - Radboud University Medical Center, Nijmegen
  - Stichting HagaZiekenhuis, The Hague
- Peru (2):
  - Hospital Militar Central Coronel Luis Arias Schreiber, Lima
  - Hospital Maria Auxiliadora, Lima
- Portugal (6):
  - Hospital de Braga, Sao Victor, Braga District
  - Hospital de Braga, Braga
  - Centro Clinico Champalimaud, Lisbon
  - Champalimaud Clinical Center, Lisbon
  - Hospital de Santa Maria - Centro Hospitalar Universitario Lisboa Norte, Lisbon
  - Centro Hospitalar Universitário de São João, Porto
- Singapore (2):
  - National Cancer Centre Singapore, Singapore
  - Raffles Hospital, Singapore
- South Korea (14):
  - National Cancer Center, Goyang-si, Gyeonggi-do
  - CHA Bundang Medical Center, CHA University, Seongnam-si, Gyeonggi-do
  - Seoul National University Bundang Hospital, Seongnam-si, Gyeonggi-do
  - The Catholic University of Korea, St. Vincent's Hospital, Suwon, Gyeonggi-do
  - Jeonbuk National University Hospital, Jeonju, Jeollabuk-do
  - Chonnam National University Hwasun Hospital, Hwasun-gun, Jeollanam-do
  - Wonkwang University Hospital, Iksan-si, Jeonlabuk-do
  - Inje University Haeundae Paik Hospital, Busan
  - Kosin University Gospel Hospital, Busan
  - Gachon University Gil Medical Center, Incheon
  - Korea University Anam Hospital, Seoul
  - Kangbuk Samsung Hospital, Seoul
  - Severance Hospital Yonsei University Health System, Seoul
  - Asan Medical Center - Oncology, Seoul
- Spain (33):
  - Complejo Hospitalario Universitario de Santiago, Santiago de Compostela, A Coruna
  - Farmacia Oncologica - Unidad de Ensayos Clinicos, Santiago de Compostela, A Coruna
  - Institut Catala d' Oncologia de Badalona - Hospital Universitari Germans Trias i Pujos, Badalona, Barcelona
  - Institut Catala d'Oncologia Badalona (ICO Badalona) - Hospital Universitari Germans Trias i Pujol, Badalona, Barcelona
  - Institut Catala d'Oncologia - Hospital Duran i Reynals (ICO L'Hospitalet), L'Hospitalet de Llobregat, Barcelona
  - Hospital de Cruzes, Barakaldo, Bizkaia
  - Hospital Universitario Marques de Valdecilla, Santander, Cantabria
  - Hospital Universitario Puerta de Hierro - Majadahonda, Majadahonda, Madrid
  - HUB-Hospital Universitario Badajoz, Badajoz
  - Infanta Cristina Hospital, Badajoz
  - Hospital Del Mar, Barcelona
  - ASCIRES CETIR Viladomat, Barcelona
  - Hospital Universitari Vall D Hebron, Barcelona
  - Hospital Universitari Vall d'Hebron, Barcelona
  - Hospital Clinic de Barcelona, Barcelona
  - Hospital de la Santa Creu i Sant Pau- Pharmacy, Barcelona
  - Hospital de La Santa Creu i Sant Pau, Barcelona
  - Unitat d'Assajos Clinics Servei de Farmacia, L'Hospitaler de Llobregat
  - Complejo Hospitalario Universitario Insular Materno-Infantil, Las Palmas de Gran Canaria
  - Hospital Universitario Nuestra Señora del Rosario, Madrid
  - Hospital General Universitario Gregorio Maranon, Madrid
  - Clinica Fuensanta, Madrid
  - MD Anderson Cancer Center Madrid, Madrid
  - Hospital Universitario Ramon y Cajal, Madrid
  - Hospital Universitario 12 de Octubre, Madrid
  - Hospital Universitario La Paz: Servicio de Farmacia, Madrid
  - Hospital Universitario La Paz, Madrid
  - Hospital Universitario HM Sanchinarro, Madrid
  - Complejo Hospitalario Universitario de Ourense (CHOU), Ourense
  - Hospital Universitario Central de Asturias, Oviedo
  - Hospital Universitario Virgen Del Rocio, Seville
  - Consorcio Hospital General Universitario de Valencia (CHGUV), Valencia
  - Hospital Universitario Miguel Servet, Zaragoza
- Sweden (2):
  - Ryhov Hospital, Jönköping
  - Karolinska University Hospital, Stockholm
- Taiwan (16):
  - China Medical University Hospital, Taichung, Taiwan (r.o.c.)
  - Chiayi Chang Gung Memorial Hospital, Chiayi City
  - Chiayi Chang Gung Memorial Hospital, Chiayi County
  - Kaohsiung Medical University Hospital, Kaohsiung City
  - Kaohsiung Chang Gung Memorial Hospital, Kaohsiung City
  - Chang Gung Memorial Hospital Kaohsiung Branch, Kaohsiung City
  - China Medical University Hospital - Pharmacy, Taichung
  - Taichung Veterans General Hospital Clinical Trials Pharmacy, Taichung
  - Taichung Veterans General Hospital, Taichung
  - Clinical Trial Pharmacy, Department of Pharmacy, National Cheng Kung University Hospital, Tainan
  - National Cheng-Kung University Hospital, Tainan
  - Chi Mei Hospital liouying, Tainan
  - National Taiwan University Hospital, Investigational Drug Service, Taipei
  - National Taiwan University Hospital, Taipei
  - Linkou Chang Gung Memorial Hospital - Clinical Trial Pharmacy, Taoyuan
  - Linkou Chang Gung Memorial Hospital, Taoyuan
- United Kingdom (4):
  - Barts Health NHS Trust , The Royal London Hospital, London
  - Barts Health NHS Trust Saint Bartholomews Hospital, London
  - Guy's and St Thomas' NHS Foundation Trust, London
  - Guy's and St Thomas' NHS Foundation, London

IPD SHARING:
Plan to Share IPD: Yes
Pfizer will provide access to individual de-identified participant data and related study documents (e.g. protocol, Statistical Analysis Plan (SAP), Clinical Study Report (CSR)) upon request from qualified researchers, and subject to certain criteria, conditions, and exceptions. Further details on Pfizer's data sharing criteria and process for requesting access can be found at: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests.
URL: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://pmiform.com/clinical-trial-info-request?StudyID=SGNDV-001